CLINICAL TRIAL: NCT05794217
Title: A Multi-Site Leukopak Repository Providing Annotated Biospecimens for Approved Investigator-Directed Biomedical Research Initiatives
Status: Recruiting | Type: Observational
Sponsor: Sanguine Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: SAN-BB-LEUK-01
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Rare Diseases
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The studies collected biospecimens are white blood cells, specifically leukopaks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: This is a non-interventional study — This is a non-interventional study

SUMMARY:
To collect, preserve, and distribute annotated leukopak biospecimens and associated medical data to institutionally approved, investigator-directed biomedical research to discover and develop new treatments, diagnostics, and preventative methods for specific and complex conditions.

This protocol will be utilized to collect research grade products that are not meant for transfusion.

DETAILED DESCRIPTION:
This is a multi-center study, with up to 20,000 participants enrolled. Participants may complete up to two visits, a screening visit, and an apheresis visit, during their enrollment in the study.

The biospecimens collected by apheresis may be processed and stored, delivered frozen, or delivered unfrozen directly to the requesting researcher. All participant specimens, if processed, will be stored, and distributed to researchers in an anonymized fashion.

The following activities will occur during the study:

Sponsor Obtain overall study informed consent. Sanguine will implement a software-as-a-service (SaaS) provider of electronic signature technology and transaction management solutions and/or a hardcopy of the informed consent form (ICF). Participants may electronically sign the ICF and authorization of release of information using an electronic device. The Sponsor will also provide the participant the option of completing hardcopy documents if they so desire. In addition to the Principal Investigator (PI), approved study staff can also administer and sign the ICF and will address all of the participant's queries regarding the ICF and study design. The informed consent process can take place at the site location by the on-site staff. In addition to the overall study informed consent, sites may also administer their own ICF per site-specific procedures, if required.

Health information will be collected via self-report and medical record review to obtain a detailed clinical history of the subject's health. The health information includes but is not limited to demographic and lifestyle information, height and weight, current medications and comorbidities, date of diagnosis, condition-related treatment history, current disease characteristics, diagnostic reports, and family medical history.

Apheresis Center Laboratory tests, including, but not limited to, a complete blood count (CBC) and viral testing for hepatitis C, hepatitis B, and HIV, at a minimum, will be performed on all prospective donors.

Apheresis health questionnaire to identify potential health risks and risk of communicable disease.

Venous access check completed by an apheresis nurse to qualify donor as having adequate veins for successful apheresis.

Assessment performed by the apheresis collection center on the day of donation which may include (but is not limited to the following) Basic health questionnaire to assess donor suitability for apheresis Mini physical exam including vitals and hemoglobin measurement Other requirements of the apheresis center as per standard procedure Apheresis cell collection

ELIGIBILITY:
Inclusion Criteria:

* Persons deemed healthy enough for the procedure and aged 18 to 89 years at the date of informed consent.

Minimum weight of 110 lbs. Pulse greater than 50 and less than 110 beats per minute Blood Pressure diastolic greater than 50 mmHg and less than100 mmHG and systolic is greater than 90 mmHg and less than 180 mmHg Peripheral veinous access is deemed adequate for apheresis as determined by apheresis staff.

Negative for Hepatitis B, Hepatitis C, and HIV 1-2 upon testing performed within 30 days, unless specifically obtaining cell collection based upon this diagnosis.

CBC results which fall within site-specific parameters within 30 days of apheresis procedure:

The participant understands the procedures and requirements of the study by providing written informed consent, including consent for authorization for protected health information disclosure.

Exclusion Criteria:

* Persons younger than 18 years of age or older than 89 years of age at the date of informed consent.

Presenting with a history of a specific condition determined through medical evaluation to be incompatible with safely undergoing apheresis Receipt of transfusion of blood products within 30 days of the study procedure. Receipt of an investigational (unapproved) drug 30 days before the study procedure.

A confirmable diagnosis of any medical condition that would increase potential procedure risks. Such medical conditions include:

Severe or untreated cardiovascular, kidney, liver, or lung diseases which would preclude apheresis procedures; Bleeding disorders Conditions associated with chronic anemia Active systemic infection Use of ACE inhibitors unless they can safely be held for 24 hours prior to apheresis procedure Pregnancy Has donated a unit of blood within the last 2 months at the date of informed consent.

Unable to understand the procedures and requirements of the study in order to provide written informed consent, including consent for authorization for protected health information disclosure.

Requires a Legally Authorized Representative (LAR) for the study informed consent.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a multi-center study, with up to 20,000 participants enrolled. Participants may complete up to two visits, a screening visit, and an apheresis visit, during their enrollment in the study.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Leukopak | September 2022 and September 2024
  The studies collected biospecimens are white blood cells, specifically leukopaks.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanguine Biosciences, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with researchers via redacted medical records.